CLINICAL TRIAL: NCT06665802
Title: Avoidant and Restrictive Food Intake Disorders (ARFID) in Adolescence: Early Oral Development, Psychopathological Profile and Sensory Integration
Acronym: ARFIDOS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240861; 2024-A01593-44 (Other: IDRCB)
Record Dates: First submitted 2024-10-24; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Avoidant and Restrictive Food Intake Disorders
Keywords: Avoidant and Restrictive Food Intake Disorders; ARFID; Eating disorder; Adolescent; Depression; Autism; Anxiety; Sensory sensitivity
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Feeding and Eating Disorders; Depression; Autistic Disorder; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ARFID adolescents: Children between 12 and 17 years old diagnosed with ARFID less than 2 years prior
  Interventions: Behavioral: Questionnaire
- Non ARFID adolescents: Children between 12 and 17 years old with no organic or psychological illness diagnosed
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire completion

SUMMARY:
The purpose of this study is to assess if adolescents affected with Avoidant and Restrictive Food Intake Disorders (ARFID) had more frequent precocious pediatric feeding disorders before 4 years old compared to healthy adolescents.

DETAILED DESCRIPTION:
This research focuses on retrospective analysis of early pediatric feeding disorders seen for ARFID in adolescence in two departments of the DMU MEFADO.

This assessment will be implemented during a hospital visit by a questionnaire completed by the patient's parents covering the first years of the child's life in medical, behavioural and dietary terms. This questionnaire was created for this study and, therefore, is not validated for general population. The parents will also complete the Montreal Children Feeding scale based on their memories.

The Montreal Children Feeding scale is a validated parental self-questionnaire, allowing the screening of feeding and eating disorders in children under 6 years old. Since the study specific questionnaire is not validated, 60 non-ARFID controls will be included in the study for questionnaires completion. The research also focuses on the psychopathological profile of these adolescents with ARFID regarding their degree of anxiety, their degree of depression, their possible autistic traits and their sensory sensitivity. These aspects will be studied by validated self- and hetero-questionnaires standardized for these fields. The emotional expression of the parents will be assessed during a brief qualitative interview type "Five-Minute Speech Sample".

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Adolescent aged 12 to 18 (minors = 17 years 11 months)
* No opposition from parents and adolescent

For ARFID patients:

* Consulting at MDA or Necker for an ARFID diagnosed using DSM V criteria
* Whose first consultation for this disorder was less than 2 years ago

For non-ARFID patients:

* Consulting or hospitalized in orthopaedic surgery at Necker Hospital or Robert Debré Hospital for an acute traumatic reason
* Not diagnosed with a chronic illness

Exclusion Criteria:

For all patients:

- Parents and adolescents who do not speak French well enough to understand the questions on the scales and questionnaires

For ARFID patients:

- Diagnosis of autism spectrum disorder already made at the time of the consultation

For non-ARFID patients:

- Presence of a chronic organic or psychological illness, to limit the risk of including non ARFID patients at high risk of eating disorders

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents diagnosed with ARFID less than 2 years before
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of pediatric feeding disorders (PFD) | 1 day
  Determine whether adolescents recently diagnosed with ARFID have more frequent FPD before the age of 4 years compared to adolescents without ARFID by using the Montreal scale score (61 or more) and/or the specific study questionnaire (at least 4 positive answers)

SECONDARY OUTCOMES:
Severity of eating disorders on growth consequences in ARFID adolescents | 1 day
  Evaluation of growth effects of ARFID by measuring the Z score and Tanner stage.
Sensory profile in ARFID adolescents | 1 day
  Determine whether adolescents recently diagnosed with ARFID have more frequent hypersensoring or hyposensoring traits compared to adolescents without ARFID by using Sensoring Processing Scale Inventory (SPSI)
Anxiety in ARFID adolescents | 1 day
  Determine whether adolescents recently diagnosed with ARFID have more frequent anxiety compared to adolescents without ARFID by using the GAD-7 scale (score of 5 or more)
Depression in ARFID adolescents | 1 day
  Determine whether adolescents recently diagnosed with ARFID have more frequent depression compared to adolescents without ARFID by using the ADRS (Adolescent Depression Rating Sclale) (score of 4 or more)
Autistic traits in ARFID adolescents | 1 day
  Determine whether adolescents recently diagnosed with ARFID have more frequent autistic traits compared to adolescents without ARFID by using the Autism Spectrum Screening Questionnaire (ASSQ) (score of 13 or more)
Parental profile in ARFID adolescents | 1 day
  Compare parent's emotional expression for adolescents recently diagnosed with ARFID to adolescents without ARFID by using the five minute speech sample.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Cochin, Paris
  - Hôpital Necker - Enfants malades, Paris
  - Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abadie V. [Diagnostic approach in oral disorder in young children]. Arch Pediatr. 2004 Jun;11(6):603-5. doi: 10.1016/j.arcped.2004.03.040. No abstract available. French. PMID 15158850
- [Background] Rein Z, Perdereau F, Curt F, Jeammet P, Fermanian J, Godart N. Expressed emotion and anorexia nervosa: the validation of the Five-Minute Speech Sample in reference to the Camberwell Family Interview. Int J Eat Disord. 2006 Apr;39(3):217-23. doi: 10.1002/eat.20245. PMID 16511834
- [Background] Goday PS, Huh SY, Silverman A, Lukens CT, Dodrill P, Cohen SS, Delaney AL, Feuling MB, Noel RJ, Gisel E, Kenzer A, Kessler DB, Kraus de Camargo O, Browne J, Phalen JA. Pediatric Feeding Disorder: Consensus Definition and Conceptual Framework. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):124-129. doi: 10.1097/MPG.0000000000002188. PMID 30358739
- [Background] Fisher MM, Rosen DS, Ornstein RM, Mammel KA, Katzman DK, Rome ES, Callahan ST, Malizio J, Kearney S, Walsh BT. Characteristics of avoidant/restrictive food intake disorder in children and adolescents: a "new disorder" in DSM-5. J Adolesc Health. 2014 Jul;55(1):49-52. doi: 10.1016/j.jadohealth.2013.11.013. Epub 2014 Feb 5. PMID 24506978
- [Background] Diagnosis and Statistical Manual of Mental Disorders: DSM-5. 5th ed. Washington, DC, USA: American Psychiatric Association (2013).
- [Background] Monteleone P, Di Genio M, Monteleone AM, Di Filippo C, Maj M. Investigation of factors associated to crossover from anorexia nervosa restricting type (ANR) and anorexia nervosa binge-purging type (ANBP) to bulimia nervosa and comparison of bulimia nervosa patients with or without previous ANR or ANBP. Compr Psychiatry. 2011 Jan-Feb;52(1):56-62. doi: 10.1016/j.comppsych.2010.05.002. Epub 2010 Jul 1. PMID 21220066
- [Background] Galmiche M, Dechelotte P, Lambert G, Tavolacci MP. Prevalence of eating disorders over the 2000-2018 period: a systematic literature review. Am J Clin Nutr. 2019 May 1;109(5):1402-1413. doi: 10.1093/ajcn/nqy342. PMID 31051507
- See also: website for parents and professionals about pediatric feeding disorders — http://inforalite.fr
- See also: website about eating behaviour of adolescents especially anorexia and bulimia nervosa — https://ffab.fr/